CLINICAL TRIAL: NCT03920319
Title: Effect of Bupropion Treatment on Brain Activation Induced by Cigarette-Related Cues in Smokers
Brief Title: Bupropion and Cigarette-Related Cues in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Brody011
Record Dates: First submitted 2019-04-13; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Smoking; Smoking, Tobacco
MeSH Terms: conditions — Smoking; Tobacco Smoking | interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, before-after controlled trial
Who Masked: Participant, Care Provider
Masking Description: Matching placebo pills
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupropion (Experimental): Participants assigned to 150mg of bupropion daily for the first 3 days, followed by titration up to 2 pills daily, separated by 8 hours, for the remaining 8 weeks of treatment.
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Participants assigned to pill placebo daily for the first 3 days, followed by titration up to 2 pills daily, separated by 8 hours, for the remaining 8 weeks of treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion — Bupropion 150 mg sustained release
  Other Names: bupropion HCl; Wellbutrin
  Arms: Bupropion
Other: Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, before-after controlled trial to assess changes in regional brain activation in response to cigarette-related cues from before to after treatment with bupropion (vs placebo).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-seeking cigarette smoker
* Meet DSM-IV criteria for nicotine dependence
* Negative result on urine test for drug use during screening

Exclusion Criteria:

* History of any Axis I psychiatric diagnosis other than nicotine dependence
* Medical conditions that might affect brain function
* Current use of medications that could alter brain function
* Pregnancy
* Current illicit drug use other than occasional use of marijuana

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2005-12-31 (Actual)

PRIMARY OUTCOMES:
Craving ratings | 8 weeks
  Participants were instructed to respond from 1 (definitely not) to 5 (definitely) on the question, "I crave a cigarette right now", after viewing video cues.

SECONDARY OUTCOMES:
Exhaled carbon monoxide (CO) | 8 weeks
  Participants were asked to hold their breath for as long as possible, ideally 15 seconds, then to breathe out slowly into the mouthpiece of a CO monitor, aiming to empty the lungs completely.
Cigarettes per day | 8 weeks
  Self-reported number of cigarettes smoked daily during the past 7 days [??]
Fagerström Test for Nicotine Dependence (FTND) | 8 weeks
  The FTND contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. The yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.

IPD SHARING:
Plan to Share IPD: No